CLINICAL TRIAL: NCT01357837
Title: A Randomized 4 Week Phase IIa Trial Evaluating the Efficacy, Safety, and Tolerability of GRT6005, a New Centrally Acting Analgesic, in Subjects With Moderate to Severe Pain Due to Osteoarthritis (OA) of the Knee
Brief Title: Assessment of GRT6005 in Painful Osteoarthritis of the Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tris Pharma, Inc. (Industry)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 116918; 2010-022556-23 (EudraCT Number); KF6005/03 (Other: Sponsor)
Record Dates: First submitted 2011-05-19; First posted 2011-05-23 (Estimated); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Osteoarthritis of the Knee
Keywords: Osteoarthritis, knee; Analgesia; Pain; Painful
MeSH Terms: conditions — Osteoarthritis, Knee; Agnosia; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Matching Placebo (Placebo Comparator): Once daily oral administration of matching placebo for 4 weeks.
  Interventions: Drug: Matching Placebo
- 75 µg GRT6005 (Experimental): Once daily oral administration of GRT6005 for 4 weeks.
  Interventions: Drug: GRT6005
- 200 µg GRT6005 (Experimental): Once daily oral administration of GRT6005 for 4 weeks.
  Interventions: Drug: GRT6005
- 400 µg GRT6005 (Experimental): Once daily oral administration of GRT6005 for 4 weeks.
  Interventions: Drug: GRT6005

INTERVENTIONS:
Drug: Matching Placebo — 2 capsules of matching placebo once a day, in the morning, for a total of 28 days
  Arms: Matching Placebo
Drug: GRT6005 — 2 capsules containing a total of 75 µg GRT6005 once a day, in the morning, for a total of 28 days
  Arms: 75 µg GRT6005
Drug: GRT6005 — 2 capsules containing a total of 200 µg GRT6005 once a day, in the morning, for a total of 28 days
  Arms: 200 µg GRT6005
Drug: GRT6005 — 2 capsules containing a total of 400 µg GRT6005 once a day, in the morning, for a total of 28 days
  Arms: 400 µg GRT6005

SUMMARY:
The purpose of the trial is to determine whether GRT6005 is effective in patients with pain due to osteoarthritis of the knee.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety, tolerability and efficacy of 3 doses of GRT6005 taken once daily for 4 weeks in outpatients with moderate-to-severe painful osteoarthritis of the knee.

ELIGIBILITY:
Inclusion Criteria:

* painful Osteoarthritis of the knee based on American College of Rheumatology Criteria
* signed informed consent
* on stable analgesic medications for painful osteoarthritis with regular analgesic intake for at least 3 months
* pain intensity score of 4 or greater on the 11-point numeric rating scale (where 0 indicates "no pain" and 10 indicates "pain as bad as you can imagine").

Exclusion Criteria:

* Substance Abuse
* Significant cardiac disease
* Presence of risk factors for Torsades de Pointes and chronic severe cardiac disease
* History of seizure disorder
* Chronic gastrointestinal disease
* Conditions that contribute and confound to the assessment of pain
* Surgery or painful procedure during or within 3 months of enrollment
* Cancer
* Subjects with impaired renal function
* Subjects with impaired hepatic function
* Female subjects who are breastfeeding
* History of chronic hepatitis B or C or human immunodeficiency virus infection, or presence of acute hepatitis A, B, or C within the past 3 months.
* Clinically relevant history of hypersensitivity or allergy to paracetamol, opioids or the excipients.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2011-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the pain intensity scores during the last week of the 4-week treatment period | 4 weeks

SECONDARY OUTCOMES:
Change from baseline in the Western Ontario McMaster Questionnaire (WOMAC) Global Score Assessing Pain, Disability and Joint Stiffness of the Knee Over the 4 week treatment period | 4 weeks
Change from baseline in quality of health as measured by Short Form-12 Health Survey | 4 weeks
Response measured in percentage change of pain intensity since baseline | 4 weeks
Leeds Sleep Evaluation Questionnaire to quantify subjective impressions of sleep and waking | 4 weeks
Patient's Global Impression of Change (PGIC) | 4 weeks
Clinician's Global Impression of Change (CGIC) | 4 weeks
Weekly current pain intensity changes from baseline | 4 weeks
Rescue medication use | 4 weeks
Quality of Life EuroQoL-5 Dimension score, change from baseline | 4 weeks
Clinical Opioid Withdrawal Scale | 4 weeks
Plasma concentration | 4 weeks
Discontinuation from study due to treatment related adverse events | 4 weeks
Time to withdrawal from study | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Olas, MD, Principal Investigator — Specjalistyczne Centrum Medyczne NZOZ NOWOMED,
Locations (26):
- Austria (5):
  - Site 3604, Linz
  - Site 3605, Senftenberg
  - Site 3603, Vienna
  - Site 3602, Vienna
  - Site 3601, Vienna
- Poland (11):
  - Site 3203, Bialystok
  - Site 3202, Elblag
  - Site 3208, Gdynia
  - Site 3206, Krakow
  - Site 3207, Lublin
  - Site 3210, Szczecin
  - Site 3201, Torun
  - Site 3211, Warsaw
  - Site 3204, Warsaw
  - Site 3205, Wroclaw
  - Site 3213, Włoszczowa
- Spain (10):
  - Site 3303, A Coruña
  - Site 3305, Barcelona
  - Site 3302, Barcelona
  - Site 3312, Málaga
  - Site 3308, Mérida
  - Site 3310, Oviedo
  - Site 3311, Petrel
  - Site 3304, Santiago de Compostela
  - Site 3306, Seville
  - Site 3313, Torrelavega